CLINICAL TRIAL: NCT03199781
Title: Motorized Mechanical Massage Associated With Cosmetics in Improving Body Contour and Appearance of Gynoid Lipodystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Principal Investigator, Renata Michelini Guidi, Principal Investigator, Indústria Brasileira Equipamentos Médicos - IBRAMED
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ibramed
Record Dates: First submitted 2017-05-19; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cellulitis of Leg
Keywords: cellulits of leg; Motorized power massage; massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention of mechanical massage with cosmetics (Experimental): Patients will be treated with motorized mechanical massage and associated with cosmetics with lipolytic active principle, being performed twice a week totaling 10 sessions by a dermato-functional physiotherapist.
  Interventions: Device: Motorized mechanical massage with the Dermothonus Slim® Ibramed with cosmetics

INTERVENTIONS:
Device: Motorized mechanical massage with the Dermothonus Slim® Ibramed with cosmetics — Patients will be treated with motorized mechanical massage with the Dermothonus Slim® electromedical equipment (Ibramed- Brazilian Industry of Electrical Equipment) associated with cosmetics with lipolytic active principle, being performed twice a week totaling 10 sessions by a dermato-functional physiotherapist.

SUMMARY:
PURPOSE: To evaluate the efficacy of motorized mechanical massage associated with cosmetics in improving body contour and appearance of gynoid lipodystrophy.

SUBJECTS AND METHODS: A prospective and comparative longitudinal clinical study will be performed in 30 women with localized fat and gynoid lipodystrophy. Patients will be submitted data collection and assessments and before and after treatment.

HYPOTHESES: It is expected that the patients will present improvement in the body contour and in the picture of the gynoid lipodystrophy after the association of the therapies.

STATISTICAL ANALYSIS: A descriptive analysis will be done before and after vibration-oscillatory therapy, with frequency tables for categorical and descriptive variables (mean, standard deviation, median, minimum and maximum values) for continuous or numerical variables. In order to compare the main variables between the groups and the collection times, the analysis of variance (ANOVA) for repeated measurements will be used. Tukey's test will be used to compare groups. The level of significance adopted for the statistical tests will be 5% or p <0.05.

DETAILED DESCRIPTION:
After signing the informed consent, the participants will be evaluated by two physiotherapists where the data collected will be from personal data, anthropometric and complementary diagnostic tests such as: ultrasound diagnosis in order to evaluate the thickness of the adipose tissue and Cutomiter analysis of the Viscoelasticity of the skin. Afterwards they will be divided and started the treatment with another physiotherapist who will perform the following protocol of the study: exfoliation of the skin, application of the motorized mechanical massage with the device Dermotonus Slim with 550mg of vacuum, continuous mode, for 20 minutes subdivided into region Abdominal and posterior thigh, after the end will be applied the creams for lipolytic purposes. The protocol will be performed twice a week for 1 hour each, totaling 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, over 18 years of age;
* With a body mass index up to 29.9 considered overweight;
* Carriers of GI lipodystrophy;
* Non smokers;
* That they agree to participate and sign the term of free and informed commitment - TCLE

Exclusion Criteria:

* Male gender;
* Performed esthetic treatment in the gluteal region and thighs in the last month;
* Patients with skin lesions, such as dermatitis and dermatoses;
* Patients with capillary fragility;
* Patients with acute deep vein thrombosis (DVT);
* On or near cancerous lesions;
* Patients with cardiac pacemaker or other implanted electronic device.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-08-20 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Anthropometric evaluation | Ten minutes
  BMI (kg / height m2)
Anthropometric evaluation | Ten Minutes
  Perimeter in the region to be treated in centimeters.
Evaluation of the degree of cellulite | Ten minutes
  Assessment of Gland Lipodystrophy: Cellulite Severity Scale (CSS). Photographic study.
Assessment of adipose tissue thickness | Twenty minutes
  Assessment of the thickness of the dermis or hypodermis (Ultrasound diagnosis)
Assessment of skin elasticity | Twenty minutes
  Evaluation of skin elasticity (Cutometer® MPA580)

CONTACTS AND LOCATIONS:
Overall Officials: Débora modena, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Ibramed - Indústria Brasileira de Equipamentos Médicos, Amparo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chang P, Wiseman J, Jacoby T, Salisbury AV, Ersek RA. Noninvasive mechanical body contouring: (Endermologie) a one-year clinical outcome study update. Aesthetic Plast Surg. 1998 Mar-Apr;22(2):145-53. doi: 10.1007/s002669900182. PMID 9502849
- [Result] Adcock D, Paulsen S, Jabour K, Davis S, Nanney LB, Shack RB. Analysis of the effects of deep mechanical massage in the porcine model. Plast Reconstr Surg. 2001 Jul;108(1):233-40. doi: 10.1097/00006534-200107000-00038. PMID 11420530
- [Result] Gordon C, Emiliozzi C, Zartarian M. Use of a mechanical massage technique in the treatment of fibromyalgia: a preliminary study. Arch Phys Med Rehabil. 2006 Jan;87(1):145-7. doi: 10.1016/j.apmr.2005.08.125. PMID 16401454
- [Result] Milani GB, Natal Filho A, Amado Joao SM. Correlation between lumbar lordosis angle and degree of gynoid lipodystrophy (cellulite) in asymptomatic women. Clinics (Sao Paulo). 2008 Aug;63(4):503-8. doi: 10.1590/s1807-59322008000400015. PMID 18719762